CLINICAL TRIAL: NCT07301060
Title: Optimizing a Sensor-Enabled mHealth Intervention for Adolescents With Suboptimal Asthma Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00150433; R34HL167214 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Asthma (Diagnosis)
Keywords: Asthma; Adolescent; Digital Health; mHealth
MeSH Terms: conditions — Asthma; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ReACT Intervention Arm (Experimental): In this condition, participants will receive the full ReACT behavior change intervention. They will use a sensor to passively monitor adherence, receive general asthma education, and report on their asthma symptoms. Participants will receive training in techniques of problem-solving. In addition, they will receive ongoing text messages with adherence feedback and encouragement tailored to their pattern of adherence and symptoms.
  Interventions: Behavioral: Sensor-Enabled mHealth Intervention for Adolescents with Suboptimal Asthma Control
- mHealth standard of care control (Active Comparator): In this condition participants will use a sensor to passively monitor adherence, receive general asthma education, and report on their asthma symptoms.
  Interventions: Behavioral: mHealth standard of care control condition

INTERVENTIONS:
Behavioral: Sensor-Enabled mHealth Intervention for Adolescents with Suboptimal Asthma Control — Participants assigned to ReACT will contribute passively monitored sensor data to track their adherence to their asthma regimen. They will also report on their symptoms. These data will be used to provide tailored feedback and support delivered via text message. These messages will encourage adolescents to adhere to their asthma regimen and address barriers using problem-solving skills taught to them at baseline.
  Arms: ReACT Intervention Arm
Behavioral: mHealth standard of care control condition — Participants assigned to ReACT will contribute passively monitored sensor data to track their adherence to their asthma regimen. They will also report on their symptoms. Participants will be provided with general asthma education at baseline.
  Arms: mHealth standard of care control

SUMMARY:
Asthma affects nearly 1 in 10 teenagers in the United States and can seriously impact their health and daily life. Teens are expected to manage their asthma by taking medications correctly and paying attention to symptoms, but this can be hard. Adolescents are still developing the skills needed to manage their thoughts, feelings, and behaviors, and they often receive less help from parents during this time. Because each teen struggles in different ways and at different times, they need support that is personalized and responds to what is happening in the moment.

Smartphones offer a promising way to help teens manage asthma well. However, most existing asthma apps do not use the full range of proven behavior-change strategies or adapt to what the teen is actually doing day to day. To address this gap, our team created Responsive Asthma Care for Teens (ReACT)-a system that collects data about each time an adolescent takes or misses a dose of medication and monitors symptoms. ReACT helps teens set goals, get feedback, notice barriers, and practice problem-solving skills. Early testing showed that teens liked ReACT and that it improved the skills needed for better asthma management.

In this study, the investigators will pilot test ReACT in a study with 160 teens ages 13-17 who have poorly controlled asthma. Teens will be randomly assigned to use ReACT or a comparison intervention for six months. The comparison intervention provides basic asthma education and a place to log symptoms and medication use-similar to what they might normally receive in standard care.

Investigators will look at how well the study procedures work across multiple sites and whether ReACT improves the skills that help teens manage their asthma. The investigators will also explore whether ReACT leads to better asthma control and quality of life. Teens will complete assessments at the start of the study, at three months, and at six months. The investigators will gather information through surveys and objective data such as medication use.

By the end of this project, the investigators will know whether the ReACT system and study protocol are feasible and ready for a larger clinical trial, and will have early estimates of how much ReACT may improve asthma outcomes for teens.

ELIGIBILITY:
Inclusion criteria for adolescents are: 1) they are between 13-17 years-old; 2) they have a physician-verified diagnosis of persistent asthma for at least 6 months; 3) they have suboptimal asthma control as defined by national asthma guidelines;5 4) they have a daily inhaled corticosteroid prescription that is compatible with the ReACT sensor; and 5) the adolescent-caregiver dyad speak and read English.

Exclusion criteria are: 1) the adolescent is currently involved in an asthma management intervention beyond usual care; 2) the adolescent has a comorbid chronic health condition that may impact lung function (e.g., cystic fibrosis); 3) the adolescent has significant cognitive impairment or developmental delay that interferes with study completion, and 4) the adolescent does not have their own smart phone. Consistent with national asthma guidelines, we define suboptimal as control as a score of ≤19 on the Asthma Control Test (ACT) or by endorsing one or more of the following symptoms of on >4 days in the past 2 weeks: (a) use of any short-acting beta-agonist medication, (b) experiencing asthma symptoms (i.e., wheezing, tightness of chest, coughing) during the day or night, (c) nighttime awakening due to asthma, or (d) activity limitation or school absence due to asthma.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2025-12-22 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment | 6 months
  We will compute frequency statistics to ensure we met our recruitment goal of 50% of the sample self-identifying as a racial/ethnic minority.
Retention | 6 months
  Retention will be calculated for study arms and compared to the hypothesized rate in one-sample tests. Retention rates for sex subgroups within each arm will also be examined descriptively. Consistent with evidence-based medicine recommendations for evaluating clinical trials, our criterion for success is no more than 20% attrition.
Engagement | 6 months
  Engagement will be considered a success if the intervention and control groups complete an average of 4/7 (57%) symptom monitoring messages each week.
Acceptability | 6 months
  The ReAct Satisfaction Questionnaire is an 8-item modification of the Client Satisfaction Questionnaire that assesses overall participant satisfaction with the ReACT intervention. Participants respond on a 4-point scale.
Usability | The System Usabiltity Scale is a 10-item measure scored on a 5-point Likert scale. It assesses ease of use, learnability, user conficence, system complexity, and need for technical support.
  System Usability Scale
Burden | 6 months
  We will use the Perceived Ease of Use subscale of the ITUES to measure burden. The subscale consists of 5 items.
Qualitative Acceptability | 6 months
  We will conduct qualitative interviews with 20% of participants who complete ReACT we will administer a semi-structured interview with questions about features, usability, general impressions, and solicit unstructured feedback.

SECONDARY OUTCOMES:
Asthma Control Test | Baseline, 3 months, 6 months
  The Asthma Control Test (ACT) is a brief, standardized patient-reported outcome measure used to assess current asthma control from the patient's perspective. It is widely used in clinical practice and research to monitor symptom control and guide treatment decisions.
  The ACT contains 5 items assessing:
  Frequency of shortness of breath Nighttime awakenings due to asthma Interference with daily activities Use of rescue medication Overall self-rating of asthma control Response format and scoring Each item is rated on a 5-point Likert scale Total score ranges from 5 to 25 25 = completely controlled 20-24 = well controlled <20 = not well controlled (often used as a clinical cutoff) Higher scores indicate better asthma control
Pediatric Asthma Quality of Life Questionnaire | Baseline, 3 months, 6 months
  The Pediatric Asthma Quality of Life Questionnaire (PAQLQ) is a disease-specific, patient-reported outcome measure designed to assess how asthma affects the daily functioning and well-being of children.
  The standard PAQLQ contains 23 items across three domains:
  Symptoms (10 items) Assesses the frequency and severity of asthma symptoms such as wheezing, shortness of breath, chest tightness, coughing, and nocturnal symptoms.
  Activity Limitation (5 items) Measures limitations in physical, social, and daily activities due to asthma. Three activities are individualized: each child identifies activities most affected by their asthma.
  Two items assess general activity limitations. Emotional Function (8 items) Captures emotional responses to asthma, including frustration, fear, concern, anger, or feeling different from peers.

OTHER OUTCOMES:
Adolescent Self-Regulatory Inventory | Baseline, 3-months, 6-months
  The Adolescent Self-Regulatory Inventory (ASRI) is a self-report measure of self-regulation designed to assess adolescents' capacity to plan, monitor, and control their thoughts, emotions, and behaviors across situations. It is grounded in developmental theory emphasizing the gradual maturation of executive and regulatory processes during adolescence.
  The ASRI includes 36 items organized into two higher-order dimensions:
  Short-Term Self-Regulation (STSR)
  Reflects regulation of immediate impulses and emotions, including:
  Acting without thinking Difficulty controlling anger or frustration Problems delaying gratification Long-Term Self-Regulation (LTSR)
  Reflects regulation in service of future-oriented goals, including:
  Planning ahead Persistence Working toward long-term objectives despite obstacles These dimensions capture the developmental tension in adolescence between immediate reward sensitivity and emerging executive control.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Nemours Children's Health, Jacksonville, Florida
  - University of Kanas, Lawrence, Kansas

IPD SHARING:
Plan to Share IPD: No